CLINICAL TRIAL: NCT03839966
Title: Computerized Intervention for Loneliness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Jesse Cougle, Associate Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018.25994
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Loneliness

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive one of two treatments
Who Masked: Participant
Masking Description: Participants will not know if they are receiving the active or control treatment.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Treatment (Experimental): Interpretation Bias Modification for Loneliness
  Interventions: Behavioral: Interpretation Bias Modification for Loneliness
- Control Treatment (Active Comparator): Healthy Habits Psychoeducation and Relaxation.
  Interventions: Behavioral: Healthy Habits Psychoeducation and Relaxation

INTERVENTIONS:
Behavioral: Interpretation Bias Modification for Loneliness — Participants will receive eight treatment sessions. They will be presented with ambiguous training scenarios on a computer screen. Scenarios will be presented in two discrete formats: a word-sentence relatedness task (adapted from Beard & Amir, 2008 and Beard, Weisberg, & Amir, 2011), and a sentence completion and comprehension task (adapted from paradigms used by Mathews and Mackintosh (2000), Steinman and Teachman (2010), and Beard and Amir (2008)). Both of these formats have been used to reduce maladaptive threat interpretations and increase benign interpretations.
  Arms: Active Treatment
Behavioral: Healthy Habits Psychoeducation and Relaxation — Participants will receive eight computerized sessions consisting of psychoeducation on healthy behaviors as well as relaxing video clips with pleasant music (e.g., videos of rainforests, wildlife, and space). These sessions will be matched for time with the active condition, lasting approximately 25-30 minutes each. Psychoeducation will cover the topics of exercise, diet, hygiene, social support, healthy activities, and sleep. The relaxing videos will be presented after the psycho-education in each session. At the conclusion of the study, participants will be provided with the active IBM treatment free of charge if they wish to receive it.
  Arms: Control Treatment

SUMMARY:
This study assesses whether a month long computerized interpretation bias modification intervention will reduce levels of loneliness compared to a control treatment.

DETAILED DESCRIPTION:
This study hopes to assess whether a month long interpretation bias modification intervention will reduce levels of loneliness compared to a control treatment. Participants will be randomized into an active treatment condition or a control treatment that involves a healthy living and relaxation protocol. The investigators hypothesize that participants in the IBM condition will have lower levels of negative interpretation bias and loneliness than those in the healthy habits condition at post treatment and follow up. The investigators further hypothesize that the effects of IBM on loneliness will be accounted for by changes in interpretation bias.

ELIGIBILITY:
Inclusion Criteria:

* Score of >48 on the UCLA Loneliness Scale

Exclusion Criteria:

* Concurrent psychotherapy for social anxiety or depression
* Unstable psychotropic medication status (i.e. a change within the last month)
* History of psychotic or (hypo)manic symptoms
* Alcohol or other substance abuse or dependence within the last three months
* Previous participation in a similar IBM study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
UCLA Loneliness Scale (ULS) | Change in loneliness from baseline to post treatment (4weeks) and three month follow up (16 weeks)
  A 20 item Self report scale measuring loneliness. Scales range from 0 to 60 with higher scores indicating a higher level of loneliness.

SECONDARY OUTCOMES:
Multidimensional Scale of Perceived Social Support | Change in Perceived Social Support from baseline to post treatment (4weeks) and three month follow up (16 weeks)
  Self-report scale that measures perceived levels of social support. Scores range from 12 to 84 with higher scores indicating higher levels of perceived social support. The three subscales (friends, family and significant other) all have a range of 4 to 28 with higher scores indicating higher levels of perceived social support.
Social Phobia inventory | Change in social anxiety symptoms from baseline to post treatment (4 weeks) and three month follow up (16 weeks)
  Self-report scale that measures Social anxiety symptoms. Scores range from 0 to 68 with higher scores indicating higher levels of social anxiety symptoms.
State-Trait Inventory for Cognitive and Somatic Anxiety-Trait Version (STICSA-T) | Change in overall anxiety symptoms from baseline to post treatment (4 weeks) and three month follow up (16 weeks)
  Self-report measure used to assess overall anxiety symptoms. Scores range from 21 to 84 with higher scores indicating higher levels of overall anxiety.
Center for Epidemiological Studies Depression Scale (CES-D) | Change in depression symptoms from baseline to post treatment (4 weeks) and three month follow up (16 weeks)
  Self-report measure used to assess depressive symptoms. Total scores range from 0 to 60 with higher scores indicating a higher level of depressive symptoms.
Interpersonal Needs Questionnaire (INQ) | Change in suicide vulnerability from baseline to post treatment (4 weeks) and three month follow up (16 weeks)
  Self report measure of suicide vulnerability. Total scores range from 15 to 105, with higher scores indicating a higher vulnerability for suicide.
Interpretations Questionnaire- Social Subscale (IQ-S) | Change in interpretation style from baseline to post treatment (4 weeks) and three month follow up (16 weeks)
  Self report measure of interpretation bias of ambiguous social situations. Scales range from 0-44 with higher scores indicating a higher level of negative interpretation bias in social situations.

CONTACTS AND LOCATIONS:
Locations (1):
- Florida State University, Department of Psychology, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No